CLINICAL TRIAL: NCT05089292
Title: Increasing Breast Cancer Screening in Chinese Immigrants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Lina Jandorf, Professor, Director, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: STUDY-20-01174; R21CA249261 (NIH)
Record Dates: First submitted 2021-10-15; First posted 2021-10-22 (Actual); Results first posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Screening Mammogram
Keywords: Breast cancer screening; Health education; Chinese immigrant; Health disparities
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Intervention Model Description: Pre/Post-test design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chinese Immigrants (Experimental): NYC Chinese immigrants provided with narrative breast health education
  Interventions: Behavioral: Narrative breast health education

INTERVENTIONS:
Behavioral: Narrative breast health education — Health education program utilizing narrative messages to promote breast cancer screening in Chinese immigrant women will be delivered in a group format in the community

SUMMARY:
The long-term goal of this research is to increase breast cancer screening rates in NYC Chinese immigrants. The researchers plan to accomplish this objective by developing and testing a culturally- and linguistically-adapted Witness Project program for Chinese immigrants. To inform the intervention development, the study team will identify barriers and facilitators to breast cancer screening in Chinese immigrants through individual qualitative interviews.

A total of 156 participants will be recruited during the entire study.

In Aim 1 which started in July 2021, 60 women were recruited for in-depth interviews to assess their breast cancer knowledge, perceived barriers and benefits/risks to completing mammography, perceived susceptibility to breast cancer, fatalism, screening intention, acculturation, language preference, and health literacy.

In Aim 2, 96 women will be recruited to participate in the pilot testing of the intervention. Recruitment will take place at community sites that serve Chinese immigrants in New York City. Enrollment for Aim 2 is anticipated to start in March of 2022.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 40 years of age
* female
* born in China
* read and speak Cantonese, Mandarin, or English

Exclusion Criteria:

- none

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lina Jandorf, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose. For individual participant data meta-analysis. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Results for Aim 2 of study provided. Gatekeepers and stakeholders were not enrolled.
Period: Overall Study
Arm/Group | Chinese Immigrants
Started | 99
Completed | 99
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Chinese Immigrants
Number analyzed (Participants) | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.2 (9.162)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 99
Last Mammogram [Count of Participants; unit: Participants]
  Less than 1 year | 43
  1-2 years | 21
  More than 2 years | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Scored Above 80% in the Feasibility and Acceptability Questionnaire
Description: Post-program survey to access acceptability of adapted narrative education program. Full-scale from 0% to 100%, with a higher percent indicating greater acceptability. An arbitrary cutoff value of 80% acceptance will determine the interventions' acceptability for the study.
Time Frame: immediately post presentation (presentation approximately 1 hour)
Measure: Count of Participants; unit: Participants
Arm/Group | Chinese Immigrants
Number analyzed (Participants) | 99
Participants | 99

2. Primary Outcome: Number of Participants Who Were Engaged in Program
Description: Percent of participants who showed up to the Chinese-community-based organizations and would like to participate in the program to assess engagement rate of participants
Time Frame: Baseline
Population: 107 is the number of people in the participating Chinese-community-based organizations.
Measure: Count of Participants; unit: Participants
Arm/Group | Chinese Immigrants
Number analyzed (Participants) | 107
Participants | 99

3. Secondary Outcome: Change in Breast Cancer Knowledge
Description: Pre- and post-program survey to access change in breast cancer knowledge. Each correct answer counted as 1 point, each incorrect one as 0, and skipped questions as 0. Full scale from 0-6, with a higher score indicates more knowledge.
Time Frame: baseline and 6 months post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chinese Immigrants
Number analyzed (Participants) | 99
score on a scale
  baseline | 4.33 (1.229)
  6 months post intervention | 4.89 (1.108)

4. Primary Outcome: Percentage of Community Organizations Willing to Host Program
Description: Percentage of Chinese Community-based organizations who were willing to host the program to assess feasibility. Engagement rate of Chinese-community-based organizations was used to access feasibility
Time Frame: 7 months
Measure: Number; unit: percentage of organizations
Units Other Than Participants: organizations
Arm/Group | Chinese Immigrants
Number analyzed (Participants) | 99
Number analyzed (organizations) | 32
percentage of organizations | 22

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Chinese Immigrants
All-Cause Mortality (participants affected / at risk) | 0/99
Serious Adverse Events (participants affected / at risk) | 0/99
Other Adverse Events (participants affected / at risk) | 0/99

LIMITATIONS AND CAVEATS:
The study utilized a convenience sample recruited from Chinese community-based organizations located in New York City, which may have contributed to the high percentage of insurance involvement (100%), primary care physician access (100%), and participants living in the United States for more than 20 years. Thus, the generalizability of the findings may be limited, particularly for populations with inadequate insurance coverage.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/92/NCT05089292/Prot_000.pdf
  • Informed Consent Form (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/92/NCT05089292/ICF_001.pdf